CLINICAL TRIAL: NCT03563014
Title: A Local Retrospective Observational Study to Evaluate the Treatment Patterns of mCRPC Patients in Belgium Treated With Radium-223
Acronym: BELFIGO
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20239
Record Dates: First submitted 2018-05-24; First posted 2018-06-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
Keywords: Radium-223; Metastatic castration-resistant prostate cancer; CRPC; Phase IV
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — Radium-223; radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radium-223 (Xofigo, Bay88-8223): Belgium patients with a diagnosis of mCRPC (no known visceral metastases) and who were treated with Radium-223 for this indication
  Interventions: Drug: Radium-223 (Xofigo, Bay88-8223)

INTERVENTIONS:
Drug: Radium-223 (Xofigo, Bay88-8223) — Follow the physician's prescription in routine clinical practice.

SUMMARY:
The aim of this non interventional study is to describe the proportion of Belgian mCRPC patients which were treated with 1 to 4 and 5 to 6 Radium-223 injections and the patient characteristics which are potentially associated with this proportion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of castration-resistant prostate cancer, symptomatic bone metastases and no known visceral metastases
* All consecutive patients who started Radium-223 treatment between 22 December 2014 and 01 June 2017
* Availability of medical records during the observation period (22DEC2013 - 01JUN2018)

Exclusion Criteria:

* Patients treated with Radium-223 for any reason before 22 December 2014 (for example an interventional trial)
* Patients participated in an investigational program with interventions outside of routine clinical practice during the radium-223 treatment period
* Patients received other radiopharmaceuticals for the systemic concomitant use for treatment of prostate cancer or for other use during the Radium-223 treatment period

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Belgian patients who were treated with Radium-223 for (metastatic) Castration Resistant Prostate Cancer
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with 5-6 Radium-223 injections versus 1-4 Radium-223 injections | Retrospectively analysis from 22 December 2013 to 01 June 2018

SECONDARY OUTCOMES:
The proportion of patients with 5-6 Radium-223 injections versus 1-4 Radium-223 injections by Radium-223 line of treatment (1st, 2nd and further line) | Retrospectively analysis from 22 December 2013 to 01 June 2018
The number of prior and post life prolonging systemic anti-cancer therapies will be described | Retrospectively analysis from 22 December 2013 to 01 June 2018
The characteristics of patients according to the experience of the study centers with Radium-223 | Retrospectively analysis from 22 December 2013 to 01 June 2018
  By stratification according to the number of months after the very first index date per center
The occurrence of progression post first dose of Radium-223 | Retrospectively analysis from 22 December 2013 to 01 June 2018
The occurrence of SSE related hospitalizations | Retrospectively analysis from 22 December 2013 to 01 June 2018
  SSE: Symptomatic Skeletal Events
The frequency of SSE related hospitalizations | Retrospectively analysis from 22 December 2013 to 01 June 2018
The number of discontinuation of Radium-223 | Retrospectively analysis from 22 December 2013 to 01 June 2018
The frequency of blood transfusions | Retrospectively analysis from 22 December 2013 to 01 June 2018
The overall survival in routine clinical practice | Retrospectively analysis from 22 December 2013 to 01 June 2018
The number of patients receiving first- and second-line systemic anti-cancer treatment in mCRPC | Retrospectively analysis from 22 December 2013 to 01 June 2018
The timing of progression post first dose of Radium-223 | Retrospectively analysis from 22 December 2013 to 01 June 2018
The time between last Radium-223 injection and next line of systemic anti-cancer therapy | Retrospectively analysis from 22 December 2013 to 01 June 2018
The number of patients receiving next line of systemic anti-cancer therapy | Retrospectively analysis from 22 December 2013 to 01 June 2018

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Belgium

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/